CLINICAL TRIAL: NCT05782608
Title: Efficacy of IV Ibuprofen vs Ketorolac in Controlling Post Operative Pain in Colorectal Cancer Surgeries in Obese Patient: A Randomized Double Blinded Controlled Study
Brief Title: IV Ibuprofen vs Ketorolac in Post Operative Pain in Colorectal Cancer Surgeries in Obese Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Ismail Salama, Resident of anesthesia, SICU & Pain Management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-503-2022
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Ibuprofen; Ketorolac; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ibuprofen; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (I) (Active Comparator)
  Interventions: Drug: IV ibuprofen
- group (II) (Active Comparator)
  Interventions: Drug: IV ketorolac

INTERVENTIONS:
Drug: IV ibuprofen — Group 1 will receive IV ibuprofen 400mg \ 6 hours the first dose will be administrated immediately post operative.
  Arms: group (I)
Drug: IV ketorolac — Group 2 will receive 20 mg IV ketorolac\ 6 hours the first dose will be administrated immediately post operative
  Arms: group (II)

SUMMARY:
The aim of this study is to assess the Efficacy of IV Ibuprofen and Ketorolac in the Management of Postoperative Pain in obese patients Following abdominal cancer surgery.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer in the world, after lung and breast cancer, and the 4th most reported cause of cancer death, reporting about 8.0 % of all cancer deaths According to the WHO, Egypt was ranked the 18th regarding the prevalence of obesity, and Deaths attributable to non-communicable diseases represent about 71% of the total mortality burden.Data obtained from the past 25 years suggest that the obesity is a cause of nearly 14% of cancer deaths in men and up to 20% of cancer deaths in women. Most of cases experience moderate to severe pain after colorectal surgery, So effective and individualized analgesia required after colorectal surgery, as pain response to surgery is not predicted.

Opioids are an effective analgesic for moderate to severe pain, although their efficacy is limited by adverse effects including respiratory depression, failure to reduce pain caused by tissue inflammation, nausea, emesis, drowsiness, moderate sedation, pruritus, urinary retention and ileus.

Regional anesthesia can be an alternative to opioids but according to multiple studies it was associated with technical difficulties and higher failure rates in obese patients. Ibuprofen is a nonselective inhibitor of cyclooxygenases (COX) enzymes, the inhibition ratio of COX-1 to COX 2 of Ibuprofen is 2,5:1 that has a low risk of bleeding or gastrointestinal problems, while other NSAID as for example ketorolac have an inhibition ratio of 330:1 for COX-1 to COX-2 , reason for a high risk of side effects , therefore its use is controversial in most of perioperative settings. ketorolac 10 and 20 mg and ibuprofen 400 mg have the same analgesic effect that was significant by hour 1 and persisted for 5-6 hours for each active medication.

ELIGIBILITY:
Inclusion Criteria:

* ASA class II.
* Age ≥ 18 and ≤ 65 Years.
* Patients undergoing midline abdominal incision for colorectal cancer surgery.
* Body mass index (BMI) >30 kg/m2.

Exclusion Criteria:

* Renal and hepatic insufficiency.
* Unstable cardiovascular disease.
* History of psychiatric and cognitive disorders.
* Patients allergic to medication used.
* Asthmatic patients.
* Peptic ulcer patients.
* patients on regular opioid consumption.
* History of allergy or hypersensitivity to any component of ibuprofen, other NSAIDs, opioids or COX- 2 inhibitors.
* Subjects with active significant anemia, history of asthma .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Assessment of Pain | During procedure
  Pain using visual analogue score (VAS score), Using a ruler to measure the distance in centimetres from the 'no pain marker' (or zero) to the current pain mark. This provides a pain intensity score out of 10; for example, 6 out of 10 (or 6/10).

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mahmoud Ismail Salama, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator
Supporting Information: Study Protocol
Time Frame: one year